CLINICAL TRIAL: NCT02740777
Title: Immunogenicity Study of a 2-dose Immunization Schedule of Recombinant Human Papillomavirus Virus-like Particle Vaccine (Type 16 and 18 L1 Proteins, Yeast) in Adolescent Females Aged 9 to 14 Years
Brief Title: Evaluating the 2-dose Immunization Schedule of Human Papillomavirus (HPV)-16/18 in Adolescent Females
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Zerun Biotechnology Co.,Ltd (Industry)
Collaborators: Guangxi Center for Disease Control and Prevention (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 311-HPV-1004
Record Dates: First submitted 2016-04-05; First posted 2016-04-15 (Estimated); Last update posted 2023-04-13 (Actual); Status verified 2023-04

CONDITIONS: Human Papillomavirus; Cervical Intraepithelial Neoplasia; Persistent Infection
MeSH Terms: conditions — Uterine Cervical Dysplasia; Persistent Infection

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 2-dose adolescent (Experimental): 300 adolescent girl will receive a two-dose schedule (0 day, 6 months) immunization of HPV-16/18 vaccine.
  Interventions: Biological: HPV-16/18 vaccine
- 3-dose adolescent (Experimental): 300 adolescent girl will receive a three-dose schedule (0 day, 2 months, 6 months) immunization of HPV-16/18 vaccine.
  Interventions: Biological: HPV-16/18 vaccine
- 3-dose adult (Experimental): 300 adult women will receive a three-dose schedule (0 day, 2 months, 6 months) immunization of HPV-16/18 vaccine.
  Interventions: Biological: HPV-16/18 vaccine

INTERVENTIONS:
Biological: HPV-16/18 vaccine — HPV 16 L1 virus like particles (VLP) 40μg; HPV 18 L1 VLP 20μg; Aluminium phosphate 225μg; NaCl 0.32M; Histidine buffer 10mM; Tween-80 0.01%.

SUMMARY:
To evaluate the immune non-inferiority, as measured by antibody responses, of a 2-dose immunization schedule (0, 6 months) of recombinant human papillomavirus virus-like particle vaccine (type 16 and 18 L1 proteins, yeast) (hereinafter referred as HPV-2 vaccine) in adolescent females aged 9 to 14 years in comparison to 3-dose immunization schedule (0, 2, 6 months) in young females aged 18 to 26 years.

DETAILED DESCRIPTION:
The study plans to enroll 600 adolescent females aged 9 to 14 years and 300 adult females aged 18 to 26 years. The adolescents will be divided into two cohorts, 300 each, receiving either a 2-dose (0, 6 months) immunization schedule or a 3-dose (0, 2, 6 months) immunization schedule. The adult female group will receive a 3-dose (0, 2, 6 months) immunization schedule.

Each subject shall be administrated with the studied vaccine according to either 2-dose or 3-dose schedule as above. Immediate reactions occurred during 30 minutes after each inoculation, all the local and systematic reactions occurred from 0 to 7 days after each inoculation will be recorded. All the adverse events (AEs) occurred from the first dose of administration to 1 month after the final dose of administration, as well as all the serious adverse events (SAEs) occurred from the first dose of administration to 6 months after the final dose of administration will be collected. Blood samples will be collected at day 0 (prior to immunization) , month 6 (prior to the last injection) , month 7, month 12, month 24, and month 36. All the blood samples will be tested HPV 16- and HPV 18-specific antibody titers.

ELIGIBILITY:
Inclusion Criteria:

Adult group:

* 18-26 healthy female
* enable to provide an legal identification
* have the ability to understand and sign the Informed Consent Form
* aren't pregnant and do not have pregnancy plan within the 7 months after the first injection
* used effective contraceptive method from the last menstruation, and agreed to avoid sexual activity without effective contraceptive method within the 15 days after injection

Adolescent group:

* 9-14 healthy female
* enable to provide an legal identification
* guardians have the ability to understand the Informed Consent Form, and both participant and guardian agreed to sign the Form (in case of unable to sign, the participant can use fingerprint as signature)

Exclusion Criteria:

* History of HPV infection
* Previous administration of any HPV vaccine
* History of severe allergic reaction requiring medical intervention (such as oral and throat swelling, difficulty breathing, hypotension or shock)
* History of allergic to vaccine, or to any ingredient of vaccine.
* History of epilepsy, seizures or convulsions, or family history of mental illness
* Subjects are immunocompromised or have been diagnosed as suffering from congenital or acquired immunodeficiency, HIV infection, lymphoma, leukemia, systemic lupus erythematosus (SLE), rheumatoid arthritis, juvenile rheumatoid arthritis inflammation (JRA), inflammatory bowel disease or other autoimmune diseases, administration of immunosuppressants with six months prior to the first vaccine dose.
* History of asthma, thyroidectomy, angioneurotic edema, diabetes or malignant
* Asplenia, functional asplenia, or any circumstances result of asplenia or splenectomy
* Medical diagnosis of coagulation abnormalities (eg, clotting factor deficiency, coagulation disorders, platelet anomaly) or obvious bruising or coagulation disorder
* Acute disease or chronic disease acute exacerbation 7 days prior to vaccination
* Administration of immunoglobulins and/or any blood products within 3 months, or administration of any live attenuated vaccine within 28 days, or administration of any subunit or inactivated vaccines within 14 days.
* Fever or axillary temperature> 37.0 °C before vaccination
* During menstrual period, breastfeeding, pregnancy(pregnancy test positive), or planned pregnant within 7 month
* History of hypertension, physical examination systolic blood pressure> 150mmHg and/or diastolic blood pressure> 100mmHg
* Abnormal laboratory tests parameters
* Any clinical significant disease or findings during study screening that, in the opinion of the Investigator may interfere with the study

Ages: 9 Years to 24 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 900 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2016-11 (Actual); Study Completion 2019-07 (Actual)

PRIMARY OUTCOMES:
HPV-16 and HPV-18 antibody titers (GMT) | one month after the final injection
  Compare the HPV-16 and HPV-18 specific antibody titers (GMT) between the 2-dose immunization schedule (0, 6 months) in adolescent females aged 9 to 14 years and the 3-dose immunization schedule (0, 2, 6 months) in young females aged 18 to 26 years.

SECONDARY OUTCOMES:
HPV-16 and HPV-18 antibody titers (GMT) and the seroconversion rate | 30 months after the final injection
  Compare the immunogenicity between the 2-dose (0, 6 months) and the 3-dose (0, 2, 6 months) immunization schedules in adolescent females aged 9-14 years, on the basis of: 1) antibody titers (GMT) and the seroconversion rate at one month after the final injection, 2) antibody titer persistence and 3) antibody titers at a steady status.
Local and systemic adverse events (AEs) | 6 months after the final injection
  Evaluate all local and systemic adverse events (AEs) occurred within 7 days after each inoculation, at one month and 6 month after the whole immunization

CONTACTS AND LOCATIONS:
Overall Officials: Zhaojun Mo, Principal Investigator — Guangxi Center for Disease Prevention and Control(GXCDC)
Locations (2):
- China (2):
  - Hezhou Center for Disease Prevention and Control, Hezhou, Guangxi
  - Zhongshan Center for Disease Prevention and Control, Zhongshan, Guangxi

IPD SHARING:
Plan to Share IPD: No